CLINICAL TRIAL: NCT07148427
Title: A Single-arm, Phase II Clinical Study Protocol of Lparomlimab and Tuvonralimab in Combination With Regorafenib and Chemotherapy as First-line Treatment for Locally Advanced or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Immunotherapy Combined With Anti-angiogenic Therapy and Chemotherapy for Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-GasC-QIBA-3007
Record Dates: First submitted 2025-08-24; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Gastric/Gastroesophageal Junction Adenocarcinoma
Keywords: regorafenib; chemotherapy; Iparomlimab and Tuvonralimab
MeSH Terms: interventions — regorafenib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab combination with regorafenib and chemotherapy (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab combination with regorafenib and chemotherapy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab combination with regorafenib and chemotherapy — Iparomlimab and Tuvonralimab：5mg/kg，Intravenous infusion，Q3W regorafenib：80mg，oral administration once daily from Day 1 to Day 14 chemotherapy：XELOX or SOX

SUMMARY:
A single-arm, Phase II clinical study protocol of Apatolimab Tovolimab in combination with regorafenib and chemotherapy as first-line treatment for locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in this study and has signed the informed consent form.
* Age greater than 18 years, regardless of gender.
* Histologically confirmed unresectable locally advanced or metastatic G/GEJ adenocarcinoma.
* No prior systemic treatment for unresectable locally advanced or metastatic G/GEJ adenocarcinoma. Previous neoadjuvant and/or adjuvant therapy is acceptable, but all systemic treatments must have been completed at least 6 months prior to the diagnosis of unresectable or metastatic disease.
* PD-L1 combined positive score (CPS) less than 1 as determined by tissue testing.
* At least one measurable lesion according to RECIST 1.1 criteria.
* ECOG performance status 0-1.
* Life expectancy >3 months.
* Adequate organ and marrow function:

Exclusion Criteria:

* Known HER2-positive expression (immunohistochemistry [IHC] 3+ or 2+ with a fluorescence in situ hybridization HER2:CEP17 ratio ≥2).
* Presence of other malignancies within 5 years prior to treatment, with the exception of adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, locally treated prostate cancer, and ductal carcinoma in situ (hormone therapy for non-metastatic prostate cancer or breast cancer is permitted).
* Known central nervous system metastases and/or carcinomatous meningitis.
* Patients with severe cardiac, pulmonary, hepatic, or renal dysfunction.
* Hypertension that cannot be controlled with antihypertensive medications (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg).
* History of bleeding within 4 weeks prior to screening, with any bleeding event graded as ≥3 according to CTCAE 5.0.
* Thrombotic events (arterial or venous) within 6 months prior to screening, such as cerebrovascular accident, deep vein thrombosis (excluding previously thrombosed veins deemed healed by the investigator), and pulmonary embolism.

  8. History of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.

  9. Patients who have previously received anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to approximately 2 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 2 years
Disease control rate (DCR) | Up to approximately 2 years
Duration of response (DoR) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 5 years
The incidence and severity of adverse events (AE) during the study period (Safety) | Up to approximately 2 years
  The incidence and severity of adverse events (AE) during the study period

IPD SHARING:
Plan to Share IPD: No